CLINICAL TRIAL: NCT03568305
Title: Characterization of Phenotypes of Occupational Asthma: Descriptive Study
Brief Title: Characterization of Phenotypes of Occupational Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6513
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2017-06

CONDITIONS: Occupational Asthma
Keywords: asthma; occupational asthma
MeSH Terms: conditions — Asthma, Occupational; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective of this multicenter, international study is to perform a multivariate descriptive analysis of a large population of well-defined subjects with sensitizer-induced OA ascertained by a positive SIC result in order to provide more information on the characteristics of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient
* Patient who performed a specific inhalation test with a positive result between January 2006 and December 2015.- Subject giving their consent for their participation
* Patient agreeing to use his data for research purposes

Exclusion Criteria:

* Patient objecting to the use of his data for research purposes
* Subjects under safeguard of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who performed a specific inhalation test with a positive result between january 2006 and december 2015.- Subject giving their consent for their participation
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective study to perform a multi-varied descriptive analysis of a cohort of patients with occupational asthma confirmed by a specific inhalation test | The period from from January 1st, 2006 to December 31st, 2015 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric De Blay, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de pneumologie, d'allergologie et de pathologie de l'environnement, Strasbourg, France